CLINICAL TRIAL: NCT03396159
Title: Validity of Mini Fluid Challenge to Assess Fluid Responsiveness Post Liver Transplantation
Brief Title: Validity of Mini Fluid Challenge Post Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Elayashy Mohamed Ahmed Hassan, lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N-6-2018
Record Dates: First submitted 2017-12-25; First posted 2018-01-10 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; mini fluid challenge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mini fluid challenge (Experimental): mini fluid will be given and stroke volume will be assessed before and after
  Interventions: Diagnostic Test: mini fluid challenge

INTERVENTIONS:
Diagnostic Test: mini fluid challenge — mini fluid challenge will be given to diagnose if patient is need fluid resuscitation or not

SUMMARY:
our study aim to assess the validity of using mini fluid challenge to assess the volaemic status of patients after liver transplantation

DETAILED DESCRIPTION:
After approval of institutional ethical committee and after informed patient consent, patients fulfilling criteria will be involved. Upon ICU admission, patients will be connected to full monitoring and confirming patient hemodynamic stability and no active bleeding through drains. Patients will be in supine position and baseline readings will be recorded. Fluid responsiveness will be assessed with mini fluid challenge by 150 ml of albumin 5% given over 1 minute. After fluid administration stroke volume (SV) assessed by trans thoracic echo (TTE) and other hemodynamic parameters will be recorded. Remaining 350 ml of albumin 5% will be continued over 14 minute to have total volume given 500 ml. after fluid administration SV and other parameters will be recorded. The fluid challenge will be given intravenously via a specific wide pore venous line. Fluid responsiveness will be defined as an increase in the SV by 15% after the infusion of fluid.

TT Echo Examination:

A single LVOT diameter will be measured for each patient as the distance between the inﬂection points at the base of the aortic valve cusps from the left parasternal long axis view during systole.

Assuming a circular cross section, the LVOT area will be calculated from the LVOT diameter as:

π X (LVOT diameter/ 2)2 = (LVOT diameter)2 X 0.785 Pulse wave Doppler sampling cursor will be placed in the middle of the LVOT immediately proximal to the aortic valve in 5 chamber apical view.

The sonographer manually will trace the velocity-time envelope (VTI). SV values will be calculated by multiplying VTI by cross sectional area.

ELIGIBILITY:
Inclusion Criteria:

* Patients post liver transplantation.
* ASA III- IV
* Age > 18 years

Exclusion Criteria:

* Age less than 18 years.
* Patient with fulminant liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
stroke volume | 1 minute after mini fluid administration
  assessed by trans thoracic echo

SECONDARY OUTCOMES:
heart rate | baseline 10 minutes after intensive care admission, 1 minute after mini fluid challenge and 1 minute after 500 ml of fluid administration
stroke volume | baseline 10 minutes after intensive care admission and 1 minute after 500 ml of fluid administration
  assessed by trans thoracic echo
mean arterial blood pressure | baseline 10 minutes after intensive care admission and 1 minute after 500 ml of fluid administration

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mohamed mokhtar, M.D, Study Director — kasralainy faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy Hospital , Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bechstein WO, Neuhaus P. [Bleeding problems in liver surgery and liver transplantation]. Chirurg. 2000 Apr;71(4):363-8. doi: 10.1007/s001040051066. German. PMID 10840602
- [Background] Leavy JA, Weil MH, Rackow EC. 'Lactate washout' following circulatory arrest. JAMA. 1988 Aug 5;260(5):662-4. PMID 3392792
- [Background] Kiszka-Kanowitz M, Henriksen JH, Moller S, Bendtsen F. Blood volume distribution in patients with cirrhosis: aspects of the dual-head gamma-camera technique. J Hepatol. 2001 Nov;35(5):605-12. doi: 10.1016/s0168-8278(01)00175-1. PMID 11690706
- [Background] Henriksen JH. Volume adaptation in chronic liver disease: on the static and dynamic location of water, salt, protein and red cells in cirrhosis. Scand J Clin Lab Invest. 2004;64(6):523-33. doi: 10.1080/00365510410002788. PMID 15370457
- [Derived] Mukhtar A, Awad M, Elayashy M, Hussein A, Obayah G, El Adawy A, Ahmed M, Dahab HA, Hasanin A, Elfouly A, Abdo M, Abdelaal A, Teboul JL. Validity of mini-fluid challenge for predicting fluid responsiveness following liver transplantation. BMC Anesthesiol. 2019 Apr 13;19(1):56. doi: 10.1186/s12871-019-0728-4. PMID 30987597